**Official Title:** A Multicenter, Randomized, Double-blind, Placebo-controlled clinical study to assess the efficacy and safety of Tildrakizumab in the treatment of moderate to severe plaque psoriasis of the scalp

**Document:** Statistical Analysis Plan (SAP)

NCT number: NCT03897088

**Date:** 30-Mar-2022

| Statistical Analysis Plan |
|---------------------------|
| Protocol TILD-18-20 |

Sun Pharmaceutical Industries Ltd 30-Mar-2022

Statistical Analysis Plan Study Part 1: Interim Analysis (up to Week 16) Study Part 2: Double Blind (Week 16 to Week 52) Study Part 3: Observational Safety Follow-Up (Week 52 to Week 72) A MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED CLINICAL STUDY TO ASSESS THE EFFICACY AND SAFETY OF TILDRAKIZUMAB IN THE TREATMENT OF MODERATE TO SEVERE PLAQUE PSORIASIS OF THE **SCALP** Protocol Number: TILD-18-20 IND Number: 101389 Date: 30-Mar-2022 

#### **Confidentiality Statement**

The information disclosed in connection with this Clinical Study Report is the trade secret, confidential, privileged and/or proprietary financial or commercial information of Sun Pharmaceutical Industries Ltd. and is delivered in confidence and reliance that it will not be copied or made available to any third party without the prior written consent of Sun Pharmaceutical Industries Ltd. except as may be required by federal, state, or local laws or regulations. Sun Pharmaceutical Industries Ltd. requests that this information be treated as privileged or confidential trade secret, commercial or financial information in accordance with 5 U.S. Code, sec. 552(b)(4), and that it be provided with prior written notice of any disclosure required by law.



# 95 Table of Contents

| STATI | ISTICAL ANALYSIS PLANISTICAL ANALYSIS PLAN SIGNATURESSUMMARY OF CHANGES | 2 |
|---|---|---|
| TABL | SUMMARY OF CHANGES | |
| TABL | | 1 |
| | | , |
| * | E OF CONTENTS | 4 |
| LIST ( | OF ABBREVIATIONS | |
| 1 1 | INTRODUCTION | 9 |
| 2 | STUDY OBJECTIVES | 10 |
| 2.1 | Primary Objective | 10 |
| 2.2 | Secondary Objectives | 10 |
| 2.3 | Exploratory Objective | 11 |
| 3 | OVERALL STUDY DESIGN AND TREATMENT PLAN | 11 |
| 4 5 | STATISTICAL CONSIDERATIONS OF PROTOCOL | 13 |
| 4.1 | General Statistical Consideration | 13 |
| 4.1.1 | Baseline and Study Day | 13 |
| 4.2 | Determination of Sample Size | 13 |
| 4.3 | Disposition of Subjects | 15 |
| 4.4 | Data Sets Analysed | 15 |
| 4.5 | Protocol Deviations | 16 |
| 4.6 | Demographic and Other Baseline Characteristics | 17 |
| 4.6.1 | Medical History | 18 |
| 4.7 | Prior/Concomitant Medications | 18 |
| 4.8 | Study Drug Exposure and Compliance | 19 |
| 4.9 | Efficacy Analysis | 20 |
| 4.9.1 | Primary Estimand and Intercurrent Events | 20 |
| 4.9.2 | Analysis of Efficacy Variables | 20 |
| 4.9.2.1 | Primary Efficacy Analysis | 24 |
| 4.9.2.2 | Secondary Efficacy Analysis | 25 |
| 4.9.2.3 | Exploratory Efficacy Analysis | 29 |
| 4.9.3 | Statistical / Analytical Issues | 29 |
| | LIST (1) 2 | 2.1 Primary Objective |

Body of the Data Display......46

152

153

154

155

6.1.5

6.1.6

6.1.7

6.2

| Statistical Analysis Plan Protocol TILD-18-20 | | | Sun Pharmaceutical Industries Ltd 30-Mar-2022 |
|---|---|---|---|
| 156 | 6.2.1 | Visits | 48 |
| 157 | 6.2.2 | Prior and Concomitant Medications | 48 |
| 158 | 6.2.3 | Safety | 49 |
| 159 | 6.2.4 | SAS® Procedures | 49 |
| 167 | | NDIX 1 | |
| 168 | S | SCORING | 61 |
| 169 | APPEN | NDIX 2 | DLQI |
| 170 | S | SCORING | 62 |

171

# List of Abbreviations

| Abbreviations | |
|---|---|
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ALT | Alanine transaminase |
| AST | Aspartate transaminase/serum glutamic oxaloacetic transaminase |
| BSA | Body surface area |
| CMH | Cochran-Mantel-Haenszel |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CFR | Code of Federal Regulations |
| eCRF | Electronic case report form |
| CS | Clinically significant |
| DLQI | Dermatology Life Quality Index |
| ECG | Electrocardiogram |
| ECI | Event of clinical interest |
| EoS | End of study |
| ЕоТ | End of treatment |
| ET | Early termination |
| FDA | Food & Drug Administration |
| ICH | International Conference on Harmonization |
| ICSR | Interim Clinical Study Report |
| IGA | Investigator Global Assessment |
| ITT | Intent-To-Treat |
| LOCF | last-observation-carried forward |
| M-N | Miettinen-Nurminen methodology |
| MACE | Major Adverse Cardiovascular Events |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Multiple Imputation |
| mIGA | Modified Investigator's Global Assessment |
| mITT | Modified Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| NCS | Not clinically significant |
| NRI | Non-responder imputation |
| NRS | Numeric Rating Scale |
| OC | Observed Cases |
| PASI | Psoriasis Area and Severity Index |
| PGA | Physician's Global Assessment |
| PGA-S | Physician Global Assessment of Skin |
| PN | Preferred Name |
| PP | Per Protocol |
| PSSI | Psoriasis Scalp Severity Index |
| PT | Preferred term |
| SAE | Serious adverse event |

| SAF | Safety analysis set |
|------|----------------------------------|
| SD | Standard deviation |
| SOC | System organ class |
| TEAE | Treatment-emergent adverse event |
| uITT | Uniform Intent-To-Treat |

#### 173 1 INTRODUCTION

- 174 This Statistical Analysis Plan (SAP) Amendment has been developed following the review of
- 175 Sun Pharmaceutical Industries Ltd Protocol TILD-18-20 (Version 01 Amendment 03, dated
- 176 17 Mar 2020), the corresponding case report form (CRF), SAP Version 2.0 (dated
- 177 09-June-2021).

185

- 178 This SAP describes the analysis sets and specific details for the statistical methods to be used
- for the analysis and reporting of all efficacy and safety data collected during the conduct of
- 180 Protocol TILD-18-20 during the initial blinded treatment period to Week 16, double blinded
- active treatment period from Week 16 through Week 52, and observational safety follow-up
- from Week 52 to Week 72. This SAP reflects changes to the statistical considerations in the
- protocol. When needed, this SAP supersedes the statistical considerations identified in
- Protocol TILD-18-20 and its amendments (as applicable). Where considerations are
  - substantially different, they will be identified as such in this document.
- 195 This SAP is being written with consideration of the recommendations outlined in the
- 196 International Conference on Harmonisation of Technical Requirements for Registration of
- 197 Pharmaceuticals for Human Use (ICH) E9 Guideline entitled "Guidance for Industry:
- 198 Statistical Principles for Clinical Trials", the E9 Addendum on Estimands and Sensitivity
- Analysis in Clinical Trials (R1) revision, and the most recent ICH E3 Guideline entitled,
- "Guidance for Industry: Structure and Content of Clinical Study Reports."

#### 201 2 STUDY OBJECTIVES

202 The objectives of this study are as follows:

#### 2.1 Primary Objective

203

210

211

212

218

219

220

224

225

226

227

228

- The primary efficacy objective of this study is:
- To assess the efficacy of tildrakizumab in subjects with moderate to severe scalp psoriasis, as measured by the proportion of subjects who achieve Investigator Global Assessment (IGA) mod 2011 (scalp) response from baseline at week 16. Response is defined as shown in Table 1 of Section 4.9.2 below.
- 209 The primary safety objective of this study is:
  - To assess the safety and tolerability of tildrakizumab in subjects with moderate to severe plaque psoriasis of the scalp over 52 weeks.

### 2.2 Secondary Objectives

- 213 The key secondary objectives of this study are:
- To assess the efficacy of tildrakizumab in subjects with moderate to severe plaque psoriasis of the scalp, as measured by the proportion of subjects who achieve at least 90% improvement from Baseline in the Psoriasis Scalp Severity Index (PSSI) response at Week 16 compared with placebo.
  - To assess the efficacy of tildrakizumab in subjects with moderate to severe scalp psoriasis, as measured by the proportion of subjects who achieve IGA mod 2011 (scalp) score of "clear" and "almost clear" with at least 2-point reduction from

Baseline at Week 12

 To assess the efficacy of tildrakizumab in subjects with moderate to severe plaque psoriasis of the scalp, as measured by the proportion of subjects who achieve at least 90% improvement from Baseline in the PSSI response at Week 12 compared with placebo.

233

234

235

- To assess the efficacy of tildrakizumab in subjects with moderate to severe scalp psoriasis, as measured by the proportion of subjects who achieve IGA (scalp only) of "clear" and "almost clear" with at least 2-point reduction from Baseline at Week 16.
  - To assess the efficacy of tildrakizumab in the treatment of moderate to severe plaque psoriasis of the scalp compared with placebo as measured by scalp surface area (SSA) involvement at Week 16.
- To assess the effect of tildrakizumab on IGA mod 2011 (scalp) and PSSI at other measured time points through week 52.
- To assess the effect of tildrakizumab on IGA (scalp only), Scalp Itch NRS, PASI, PGA-S (whole body), and IGA mod 2011 (whole body), at week 12 and other measured time points through Week 52.
- To assess the time to response
- To assess the efficacy of tildrakizumab in the improvement of scalp itch as measured by the proportion of subjects achieving a 4-point reduction in Scalp Itch Numeric Rating Scale (NRS) score from Baseline at Week 16 compared with placebo
- To assess the efficacy of tildrakizumab in the treatment of moderate to severe psoriasis (entire body including scalp) compared with placebo as measured by Psoriasis Area and Severity Index (PASI), IGA mod 2011 (whole body), Physician Global Assessment for skin (PGA-S) score (whole body), and total body surface area (BSA) involvement at Week 16.

### 250 **2.3** Exploratory Objective

- 251 The exploratory objective of this study is:
- To assess the effect of tildrakizumab on Quality of Life measured by: Dermatology Life Quality Index (DLQI).

### 254 3 OVERALL STUDY DESIGN AND TREATMENT PLAN

- 255 The overall study design and treatment plan are described in Sections 4.1 of Clinical Protocol
- 256 TILD-18-20 . A brief overview is included below.
- 257 This is a multicenter, randomized, double-blind, placebo-controlled Phase 3 study to assess
- 258 the efficacy and safety of tildrakizumab in the treatment of moderate to severe psoriasis of
- 259 the scalp. The study will enroll approximately 214 subjects with moderate to severe psoriasis

301

308

317

# 292 4 STATISTICAL CONSIDERATIONS OF PROTOCOL

#### 293 4.1 General Statistical Consideration

- 294 All summaries and analyses conducted will be by assigned therapy and/or combined total
- subjects. Data obtained on the eCRF and entered into the database will be provided in data
- 296 listings showing individual subject values.
- Descriptive statistics (number [n], mean, standard deviation [SD], median, first quartile [Q1],
- 298 third quartile [Q3], minimum [min], and maximum [max]) for continuous variables and
- 299 frequency distributions and percentages for discrete variables will be utilized. Categorical
- variables will be summarized by frequencies and percentages.



- All tabulations of summary statistics, graphical presentations, and statistical analyses will be
- 307 performed using SAS® Version 9.4 or higher.

### 4.1.1 Baseline and Study Day

- For purpose of the SAP, Day 1 is defined as the date of first administration of study drug.
- 310 Study day is calculated relative to the date of Day 1.
- 311 Unless otherwise specified, "Baseline" is defined as the last observed value of the parameter
- of interest prior to the first intake of study treatment (this includes unscheduled visits). For
- numerical variables, change from Baseline will be calculated as the difference between the
- 314 post-Baseline value and the corresponding Baseline value. Change from Baseline is defined
- as: post-Baseline value Baseline value. The percent change from Baseline will be calculated
- as change from Baseline divided by the Baseline value, expressed as a percentage.

#### 4.2 Determination of Sample Size

The study will randomize approximately 107 subjects per treatment arm (Total N=214)

randomization to either tildrakizumab 100 mg arm (Arm A) or placebo arm (Arm B),

387

Uniform Intent-to-Treat (uITT) Set

### 360 4.3 **Disposition of Subjects** The number and frequency of subjects who were screened, screen failures (overall and by 361 reason of screen failure), randomized, completed (overall and by each part of the study), and 362 discontinued (overall and by each part of the study) will be presented. A summary of reasons 363 364 for discontinuation will be provided. Due to the outbreak of COVID-19 pandemic, COVID-19 related subject disposition events will be further summarized per FDA Guidance on Conduct of Clinical 369 Trials of Medical Products during COVID-19 Public Health Emergency (thereinafter referred 370 to as FDA COVID-19 Guidance)<sup>a</sup>, for the following: 371 • Number of subjects discontinued from the study for reasons related to COVID-19 372 373 • Number of subjects with visits altered (e.g., remote visits) or missed due to COVID-19 374 375 • Number of subjects with any efficacy assessments not done at each visit due to 376 COVID-19 associated criteria. 378 **Data Sets Analyzed** 4.4 379 The following analysis sets will be used in the study: 380 **Intent-to-Treat (ITT) Set**: All randomized subjects who have been dispensed study 381 382 Modified Intent-to-Treat (mITT) Set:



type, either minor or major. Protocol deviations represent a failure to adhere to the clinical

study protocol. The two types of deviations are defined as:

413

414



- 436 Protocol deviations attributable to the COVID-19 pandemic regardless whether deemed
- major or minor will be provided in a separate listing if deemed necessary. Protocol
- deviations will be presented in summary tables, for IA and overall, respectively.

# 4.6 Demographic and Other Baseline Characteristics

- Demographic and baseline characteristics generally will be summarized descriptively overall
- and by treatment in the ITT, mITT, uITT, SAF, and PP analysis sets. The following
- demographic and Baseline variables will be included:
- Age (years)
- Gender
- 445 Race

439

- Ethnicity
- Prior use of TNF-alpha inhibitors (Yes/No)
- Weight (kg)
- Weight category (≤90 kg or >90 kg)
- Height (cm)
- BMI (kg/m<sup>2</sup>)
- Baseline IGA mod 2011 (scalp)
- Baseline IGA (scalp only)
- Baseline PSSI
- Baseline SSA involvement
- Baseline total BSA involvement
- Baseline IGA mod 2011 (whole body)
- Baseline PGA-S score (whole body)
- Baseline Scalp itch NRS score
- Baseline PASI score
- 463 All demographic data and baseline disease characteristics data will be listed by subject.
- 464 **4.6.1 Medical History**
- 465 Medical/surgical history and concurrent procedures will be coded using the MedDRA
- 466 (Medical Dictionary for Regulatory Activities) Version 24.0 or a more recent version and will
- be presented in a by-subject listing.
- 468 4.7 Prior/Concomitant Medications
- Prior and concomitant medications will be coded using the World Health Organization
- 470 (WHO) Drug Dictionary September 1, 2019 B3 Global. Prior medications include
- 471 medications used to treat the disease conditions and any other medications taken within 6
- 472 months prior to enrollment and stopped prior to start of treatment. Concomitant medications
- during the study are defined as any medications that are ongoing or with stop dates on or after
- date of first study medication administration.
- 475 For the determination of prior vs. concomitant medications, the following rules regarding the
- 476 stop date will be applied:
- If the stop date is missing completely, the medication is assumed to be a concomitant medication.

481

482 483

484

497

- If only year was recorded, and it is before Baseline, it is a prior medication; if year is same or after Baseline, it is assumed to be a concomitant medication.
  - If day is missing, but month and year are before Baseline, it is a prior medication; if month and year are the same as Baseline, it is assumed to be a concomitant medication; if month and year are after Baseline, it is a concomitant medication.
  - If start date is after Baseline, it is a concomitant medication regardless.



- The number and percentage of subjects taking prior medications or concomitant medications
- 492 (overall and by study parts) will be summarized by anatomical therapeutic chemical (ATC)
- level 3 and preferred name (PN) for the SAF. Although a subject may have taken two or more medications, the subject is counted only once within an ATC classification. The same subject
- 495 may contribute to two or more PTs in the same classification. All prior and concomitant
- 496 medications will be listed by subject.

# 4.8 Study Drug Exposure and Compliance

- 498 Study drug exposure will be evaluated using total number of doses administered for the entire
- 499 treatment period, and for Part 1 at interim analysis and later, Part 2

separately for final analysis. Number and percent of doses

- administered per subject and number of subjects with dose administered at each scheduled
- visit will be summarized with descriptive statistics by treatment arm (Part 1 only) and in total
- using the Safety Analysis Set.



- The study medication was originally designed to be administered at the study center by
- trained staff; however, due to the outbreak of the COVID-19 pandemic, eligible and trained
- subjects could self-administer study medication during modified remote study visits.
- 511 Self-administered study doses will be indicated in a listing.

All study drug administration data will be listed by subject.

### 4.9 Efficacy Analysis

513

514

### 4.9.1 Primary Estimand and Intercurrent Events

The primary estimand for this study is based on composite strategy approach.

## 529 **4.9.2 Analysis of Efficacy Variables**

- 530 Efficacy endpoints will be summarized descriptively by randomized treatment and by visit
- for subjects within ITT, mITT, and uITT Sets as per the specifications below. The mITT will
- be considered as the primary population for primary efficacy analysis and the uITT and PP
- Sets as supportive; the ITT will be considered as the primary population for key secondary
- and all other efficacy endpoint analysis. The mITT and uITT Sets will be considered as the
- sensitivity analysis populations for primary efficacy analyses. Subgroup analyses
- incorporating multiple definitions of response may also be performed if sufficient subjects are
- identified to contribute to such analyses.

| Protocol TILD-18-20 | 30-Mar-2022 |
|---------------------|-------------|

Sun Pharmaceutical Industries Ltd

Statistical Analysis Plan



Sun Pharmaceutical Industries Ltd

594 These key secondary endpoints will be included in multiplicity adjustments. 595 Other secondary endpoints are: Mean percentage change in PSSI score from Baseline to Week 16 596 597 The proportion of subjects achieving PSSI 75 at Week 16 599 The proportion of subjects achieving PSSI 100 at Week 16. 600 to 100%. 605 Mean percentage change in scalp surface area involvement from Baseline to Week 16. 607 608 Time to achieving IGA mod 2011 (scalp) response during the 16-week placebo-controlled 609 610

- treatment period, defined as time in days from Baseline to first achieving a score of "clear" or "almost clear" with at least a 2-point reduction from Baseline through Week 16. Subjects who have not achieved IGA mod 2011 (scalp) response by the last visit or
- 611 Week 16 will be censored at their last available assessment or Week 16 assessment, 612 whichever is later. 613
- 614 • Time to achieving PSSI 75 during the 16-week placebo-controlled treatment period, defined as time in days from Baseline to first achieving PSSI 75. Subjects who have 615 616 not achieved PSSI 75 by the last visit or Week 16 will be censored at their last available assessment or Week 16, whichever is later. 617
- The proportion of subjects decrease in Scalp itch NRS score from 618 Baseline at Week 16, assessed among subjects with Baseline Scalp Itch NRS 619
- The Scalp itch NRS is a self-administered, single item questionnaire with response 620 options from 0=No Itch to 10=Worst itch imaginable. 621
- The proportion of subjects achieving PASI 75, PASI 90, and PASI 100 622 at Week 16. Detailed PASI scoring 624 algorithms are provided in Appendix 1 PASI Scoring.



683

684

IGA (scalp only)

Scalp Itch NRS

# 712 **4.9.3 Statistical / Analytical Issues**

# 717 4.9.3.2 Handling of Dropouts or Missing Data

Data from subjects who withdraw from the study, including AEs and any follow-up, will be included in the analyses as applicable.







Sun Pharmaceutical Industries Ltd 30-Mar-2022



### 795 4.9.3.4 Multicenter Studies

Descriptive summaries of the primary and key secondary efficacy endpoints will be presented for each individual study center to evaluate potential heterogeneity across sites.





834 Several occurrences of the same AE in one subject will be counted once at the worst severity

835 grade.

The relationship of each AE to the study drug will be grouped as related (definitely, probably,

possibly related) or unrelated (unlikely to be related, unrelated). Several occurrences of the

same AE in one subject will be counted once and the one with the closest relationship to

study medication will be counted. If an AE is missing the relationship to study medication,

the event will be assumed to be related to study drug for analysis and summarization.



Non-TEAEs will be listed only and will not be included for analysis and summarization.

All AEs will be presented in a by-treatment and by-subject listing, detailing the verbatim

850 term, SOC, PT, application site reaction or not, related to study indication or not, start date,

stop date, time since most recent dose of IP, severity, outcome, relationship to study drug,

action taken regarding study drug, action taken to treat AE, seriousness and criteria for

seriousness. Serious AEs (SAEs) and TEAEs leading to study medication discontinuation,

AEs of Special Interest (AESI), and events of clinical interest (ECI) will also be presented in

separate listings.

An AE profile for the Safety Analysis Set will be provided for Part 1, Parts 2 and 3, and

overall, which summarizes the subject incidence, by treatment received for the following

858 information:

865

866

859 • Any TEAEs;

• Non-TEAEs;

• Drug-related TEAEs;

• Any TEAEs with an outcome of death;

• Treatment-emergent SAEs;

• Drug-related treatment-emergent SAEs;

• TEAEs leading to discontinuation of study medication;

• Drug-related TEAEs leading to discontinuation of study medication;

867

868

869

872

873

• Any AEs of special interest, including:

- Injection site reactions
- Severe infections
- o Malignancies (excluding carcinoma in situ of the cervix).
- 871 o Non-melanoma skin cancer
  - Melanoma skin cancer
    - o Major Adverse Cardiovascular Events (MACE)
- o Study treatment-related hypersensitivity reactions.



The number and percentage of subjects with TEAEs will be summarized for each treatment

arm and/or in total by SOC and PT. Drug-related TEAEs, TEAEs leading to discontinuation

of study drug, drug-related TEAEs leading to discontinuation of study drug, treatment-

894 emergent SAEs, and drug-related treatment-emergent SAEs will be summarized in the same

manner. For these summaries, subjects with multiple AEs will be counted only once per SOC

896 and PT.

897 TEAEs by maximum severity and TEAEs by relationship to study treatment, and commonly

occurring TEAEs, i.e., those that occur in of the subjects in either treatment arm,

will be summarized by SOC and PT by treatment received in Part 1, Parts 2 and 3, and

900 overall.

Injection site reactions will be described in a by-subject listing and may be summarized

902 separately if deemed necessary.
903 COVID-19 related adverse events may also be summarized separately if deemed necessary.

#### 4.10.2 **Clinical Laboratory Evaluation**

905 Absolute values and changes from Baseline of clinical laboratory data (hematology, 906 chemistry, continuous urinalysis parameter and lipids) will be summarized with descriptive 907



All clinical laboratory data relevant to the reporting period 912 will be

listed by subject. Values outside the normal ranges will be flagged. Flags will describe 913

914 direction relative to normal range in relevant parameters.

#### 915 **Vital Signs** 4.10.3

904

916 Vital signs measurements including temperature, pulse rate, systolic blood pressure, and 917 diastolic blood pressure, respiratory rate at each scheduled visit and changes from baseline during the treatment period will be summarized by treatment arm. Vital signs will also be 918 919 presented in a shift table displaying the cross tabulation of the Baseline result category versus

920 the result of the post-treatment period at each scheduled visit. The categories of each vital

921 sign parameters are as below:



# 923 4.10.4 12-Lead Electrocardiogram (ECG)

The ECG measurements at each scheduled visit

and change from baseline

- during the treatment period will be summarized by treatment arm.
- All ECG measurements and the overall interpretation will be listed by subject

## 930 4.10.5 Physical Examinations

- The frequency of subjects with abnormal evaluations of body system findings for physical
- examinations will be summarized by visit and treatment group; abnormal physical
- examination findings will also be presented in a by-subject listing.

#### 934 4.10.6 Performance Status

935 Not applicable.

944

## 936 4.10.7 Other Safety Parameters

- 937 The subjects will be assessed for suicidal ideation and behavior using Columbia-Suicide
- 938 Severity Rating Scale (C-SSRS) at screening, baseline and each subsequent visit. C-SSRS
- ontains two categories: (1) Suicidal Ideation (questions 1-5), most severe ideation will also be
- ollected; (2) Suicidal behavior (questions 6-10).
- The following outcomes are C-SSRS categories and have binary responses (yes/no). The
- 942 categories listed below have been re-ordered from the actual scale in an increasing order of
- severity from 1 to 10 to facilitate the definitions of the comparative endpoints.

#### Table 2 C-SSRS Outcomes

# Categories Suicidal Ideation (1-5) 1 – Wish to be dead 2 – Non-specific active suicidal thoughts 3 – Active suicidal ideation with any methods (not plan) without intent to act 4 – Active suicidal ideation with some intent to act, without specific plan 5 – Active suicidal ideation with specific plan and intent

| Categories |
|----------------------------------|
| Suicidal behavior (6-10) |
| 6 – Preparatory acts or behavior |
| 7 – Aborted attempt |
| 8 – Interrupted attempt |
| Suicidal acts (9-10) |
| 9 – Non-fatal suicide attempt |
| 10 – Completed suicide |

- The following are numerical scores derived from the above C-SSRS categories.
  - Suicidal Ideation Score: The maximum suicidal ideation category (1-5 on the C-SSRS) present at the assessment. Assign a score of 0 if no ideation is present.
    - Suicidal Behavior Score: The maximum suicidal behavior category (6-10 on the C-SSRS) present at the assessment. Assign a score of 0 if no behavior is present.
    - Suicidal Ideation or Behavior Score: The maximum suicidal ideation or behavior category (1-10 on the C-SSRS) present at the assessment. Assign a score of 0 if no ideation or behavior is present.
- 953 Subjects are also classified into two risk levels:
  - Intermediate risk level is indicated by a response of "yes" to Questions 1 to 3 and the absence of a "yes" response to Questions 4 and 5.
  - High risk level is indicated by a response of "yes" to Questions 4 or 5 in the suicidal ideation section, or any positive response in the behavioral section of the C-SSRS.
- Change in binary response to the questions from no to yes in any questions will be summarized
- in a shift table describing baseline vs post-baseline per visit, and worst post-baseline overall.
- Categorical scores will be analyzed similarly. C-SSRS risk levels are also summarized by visit.
- Results from the C-SSRS will be listed by subject. Results to Week 16 will be described in the
- Part 1 interim analysis, and overall results to Week 52 and 72 will be described in the final
- 963 analysis.

946

947

948 949

950

951

952

954

955

956

957

964

## 4.11 Sensitivity and Subgroup Analyses

- Sensitivity and subgroup analyses will be performed to confirm the robustness of primary
- analysis results.



COVID-19 impacted subjects will be identified from study tracking documentation and event-level impacts will be integrated to the EDC. Events that exceed 5% subject-level incidence of

1022

1023

the relevant analysis set will be used to exclude affected subjects from the analysis sets defined 1024 1025 for sensitivity analyses. Events that do and do not exceed a 5% subject-level incidence of the 1026 relevant analysis set will be presented using descriptive statistics for the incidence of subject-1027 level impacts via sensitivity analyses. 1028 See also Section 4.3 for presentation of COVID-19 pandemic related subject disposition. 1029 4.13 Changes from Planned Analyses in the Protocol 1030 The following changes or additions to the planned analyses described in the study protocol 1031 are noted: 1032 In Section 4.2 Determination of Sample Size, the assumption has been corrected from 1033 the protocol 'continuity-corrected Z-test with unpooled variances' to use 'continuity-1034 corrected Z-test with *pooled* variances', as a technical correction. 1035 The protocol defines an Intent-to-Treat (ITT) Set (all randomized subjects who have 1036 received at least one dose of study treatment) as the primary analysis population. The SAP further defines a modified Intent-to-Treat (mITT) Set (all randomized subjects 1037 1038 who have been dispensed dose of study treatment as the primary analysis 1039 population for the primary efficacy endpoint 1040 The SAP also further defines the uniform Intent-to-Treat (uITT) Set as the supportive 1041 analysis population for the primary efficacy endpoint. 1042 1046 Prior versions of the SAP have included an analysis of IGA (scalp only) in the ITT 1047 Set among subjects enrolled under the original protocol. This is no longer considered 1048 determinative for evaluating the effect of therapy in the indication of moderate to 1049 severe scalp psoriasis and so the analysis is moved to the 'Other Secondary' section. 1050



Sun Pharmaceutical Industries Ltd 30-Mar-2022



| | Statistical Analysis Plan Protocol TILD-18-20 Sun Pharmaceutical Industries Ltd 30-Mar-2022 |
|---|---|
| 1085 | o 4.9.1 Primary Estimand and Intercurrent Events, |
| 1086 | o 4.12 COVID-19 Pandemic Impacted Subject Assessments |
| 1087 | Section 4.9.6 describes by-subject displays |
| 1088 | Section 6.2.1 describes COVID-19 impacts to Visits |
| 1089 | Section 6.2.4 describes SAS® Procedures for M-N methodology implementation |



#### 1105 6 PROGRAMMING CONSIDERATIONS

- All tables, data listings, figures (TLFs), and statistical analyses will be generated using SAS®
- 1107 Version 9.4 or above. Generated outputs will adhere to the following specifications.

# 1108 **6.1** Table, Listing, and Figure Format

#### 1109 **6.1.1 General**

- 1110 1) All TLFs will be produced in landscape format.
- 1111 2) All TLFs will be produced using the Courier New font, size 8.
- The data displays for all TLFs will have a 1.5-inch binding margin on top of a landscape oriented page and a minimum 1-inch margin on the other 3 sides.
- 4) Headers and footers for figures will be in Courier New font, size 8.
- 1115 5) Legends will be used for all figures with more than 1 variable, group, or item displayed.
- 1117 6) TLFs will be in black and white (no color).
- 7) Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text, will not be used in the TLFs. On some occasions, superscripts 1, 2, or 3 may be used (see below).
  - 8) Only standard keyboard characters will be used in the TLFs. Special characters, such as non-printable control characters, printer-specific, or font-specific characters, will not be used. Hexadecimal-derived characters will be used, where possible, if they are appropriate to help display math symbols (e.g., µ). Certain superscripts (e.g., cm²) will be employed on a case-by-case basis.
  - 9) Mixed case will be used for all titles, footnotes, column headers, and programmer-supplied formats.

#### 1128 **6.1.2** Headers

1121

1122

1123

1124 1125

1126

1127

- 1) All output should have the following header at the top of the page:
- 1130 Sun Pharmaceutical Industries Ltd Status Draft/Final Page n of N
- 1131 Study: TILD-18-20 Interim/Final Analysis
- All output should have page number. TLFs should be internally paginated in relation to the
- total length (i.e., the page number should appear sequentially as page n of N, where N is the
- total number of pages in the table, listing or figure).

## 1135 **6.1.3 Display Titles**

Each TLF should be identified by a numeral, and the designation (i.e.,

| 1137<br>1138<br>1139<br>1140<br>1141<br>1142<br>1143 | 1) | Table 1) should be centered above the title. A decimal system (Table 14.x.y.z, Figure 14.x.y.z, and Listing 16.2.x.y) should be used to identify TLFs with related contents. The title is centered in initial capital characters. The analysis set should be identified on the line immediately following the title. The title and table designation are single spaced. A solid line spanning the margins will separate the display titles from the column headers. There will be 1 blank line between the last title and the solid line. |
|---|---|---|
| 1143 | | Table 14.x.y.z First Line of Title |
| 1145 | | Second Line of Title if Needed |
| 1146 | | FAS |
| 1147 | 6.1.4 | Column Headers |
| 1148<br>1149 | 1) | Column headings should be displayed immediately below the solid line described above in initial upper-case characters. |
| 1150 | 2) | For numeric variables, include "unit" in column or row heading when appropriate. |
| 1151<br>1152<br>1153 | 3) | Analysis set sizes will be presented for each treatment group in the column heading as (N=xx) (or in the row headings if applicable). This is distinct from the 'n' used for the descriptive statistics representing the number of subjects in the analysis set. |
| 1154 | 4) | The order of treatments in the tables and listings will be: Placebo and Tildrakizumab |

1156

1159

1160

1161

1162

1163

1166

1167

1168 1169

1170

1171

1172

1173

1174 1175

# 6.1.5 Body of the Data Display

- 1) Listings data will be sorted for presentation in order of treatment groups as above, subject ID, collection day, and collection time.
  - 2) If the categories of a parameter are ordered, then all categories between the maximum and minimum category should be presented in the table, even if n=0 for all treatment groups in a given category that is between the minimum and maximum level for that parameter. For example, the frequency distribution for symptom severity would appear as:

| Severity Rating | n |
|-----------------|---|
| severe | 0 |
| moderate | 8 |
| mild | 3 |

Where percentages are presented in these tables, any counts of 0 will be presented as 0 and not as 0 (0%).

- 3) If the categories are not ordered (e.g., Medical History, Reasons for Discontinuation from the Study, etc.), then only those categories for which there is at least 1 subject represented in 1 or more groups should be included.
- 4) An Unknown or Missing category for categorical summarization should be added to any parameter for which information is not available for 1 or more subjects.
- 5) Unless otherwise specified, the estimated mean and median for a set of values should be printed out to 1 more significant digit than the original values, and standard deviations should be printed out to 2 more significant digits than the original values. The minimum and maximum should report the same significant digits as the original values. For example, for systolic blood pressure:

| n | XX |
|--------|------------|
| Mean | XXX.X |
| SD | X.XX |
| Median | XXX.X |
| Range | (XXX, XXX) |

1176

1177

1178

11791180

1181

11821183

1184

1185

- 6) All p-values should be output in the format: "0.xxxxx", where xxx is the value rounded to 5 decimal places. Any p-value less than 0.00001 will be presented as <0.00001.
- 7) Data in columns of a table should be formatted as follows:
  - alphanumeric values are left-justified;
    - whole numbers (e.g., counts) are right-justified; and
- numbers containing fractional portions are decimal aligned.
- 8) Percentage values should be printed with 1 digit to the right of the decimal point in parentheses set 1 space after the count (e.g., 7 (12.8%), 13 (5.4%)). Less-than-signs

1189

1190

1191

1192

1193 1194

1195

1196 1197

1198

1199

1200

1201

1202 1203

1204

1205

1206

1207

1208 1209

1210

1211

1212

1218

1219

1220

- "<0.1%" should be printed when values are >0.0% and <0.1% (not 0.0%). Unless otherwise noted, for all percentages, the number of subjects in the analysis set for the treatment group who have an observation will be the denominator.
  - 9) Tabular display of data for prior / concomitant medications, and all tabular displays of adverse event data should be presented by the body system, drug class, or SOC with the highest occurrence in the active treatment group in decreasing order. Within the body system, drug class and SOC, medical history (by PT), drugs (by ATC3 code), and adverse events (by PT) should be displayed in decreasing order. If incidence for more than 1 term is identical, they should then be sorted alphabetically.
  - 10) Missing data should be represented on subject listings as either a hyphen ("-") with a corresponding footnote ("- = unknown or not evaluated"), or as "N/A", with the footnote "N/A = not applicable", whichever is appropriate. For summary tables, missing descriptive statistics or p-values due to non-estimability should be reported as "-" with a corresponding footnote ("- = not estimable")..
  - 11) Date should be printed in ISO date format ("yyyy-mm-dd": 2000-07-01). Missing portions of dates should be represented on subject listings as partial dates (2000-07). Dates that are missing because they are not applicable for the subject are output as "N/A", unless otherwise specified.
  - 12) All observed time values must be presented using a 24-hour clock HH:MM:SS format (e.g., 01:35:45, or 11:26). Time will only be reported if it was measured as part of the study.

## 6.1.6 Demographics and Baseline Characteristics

- 1) Age = (Date of informed consent Date of birth + 1) / 365.25 and truncated to complete years.
- 2) Conversion factors and calculations for height, weight, and BMI:
  - Height (in cm) = height (in inches) \* 2.54
  - Weight (in kg) = weight (in lbs) \* 0.4536
- 1213 BMI  $(kg/m^2) = Weight(kg)/[Height(m)^2]$
- 1214 3) The value of XX (e.g. age or day of assessment) will be calculated relative to a reference time point X (e.g. time of enrollment/first dose). If reference day/month is missing, the first day of the month/year will be used to create a SAS® date for variables 'Date of X'.

# 6.1.7 Footnotes

- 1) A solid line spanning the width between the left and right margins will separate the body of the data display from the footnotes.
- 2) All footnotes will be left justified with single-line spacing immediately below the solid line underneath the data display.

- 3) Footnotes should always begin with "Note:" if an informational footnote, or asterisks and other non-numeric symbols if an annotated footnote. Each new footnote starts on a new line.
  - 4) Footnotes will be present on the page where they are first referenced and thereafter on each page of the table, unless the footnote is specific only to certain pages. Subject specific footnotes should be avoided.
  - 5) Footnotes will be used sparingly and must add value to the table, figure, or data listing. If more than 4 footnotes are planned, then a cover page may be used to display footnotes, and only those essential to comprehension of the data will be repeated on each page. Footnotes should not repeat definitions already provided in the SAP.
  - 6) The last line of the footnote section will be a standard source line that indicates the data source called in by the program, the name of the program used to produce the data display, and the listing source (i.e., 'Data source: xyzabc.sas7bdat Program source: myprogram.sas Listing source: 16.x.y.z').

# 6.2 Data-Handling Rules

- 1238 This section describes naming conventions and rules for calculations that would be common
- to all applicable tables. Some rules specific to a table can be found in the relevant mock-ups.

#### 1240 **6.2.1** Visits

1226

1227

1228

1229

1230

1231

1232

1233

1234

12351236

1237

1245

1246

1249

1250 1251

12521253

1254

1255

1256 1257

1258

1259

- 1) Relative Study Day: The first day of treatment is Day 1. A minus (-) sign indicates days prior to the start of treatment (e.g., Day -5 represents 5 days before start of therapy. There is no Day 0. The relative study day for a specific post-baseline visit is calculated as (Visit Date Date of First Dose +1).
  - 2) Baseline: Evaluation taken on baseline visit or the last available evaluation prior to the first dose of study drug if the former is missing.
- 1247 3) COVID-19 affected week 16 visit: by-subject listing will show imputed and modeled results. See Section 4.11 for additional details.

## 6.2.2 Prior and Concomitant Medications

- 1) Prior and concomitant medications will be coded and classified using the treatment start and stop dates relative to date of first study medication. The specific dictionary version will be provided in the actual tables/listings.
- 2) Counting rules for prior/concomitant medications: Prior medications refer to all medications that were taken within 6 months prior to enrollment and stopped prior to start of treatment. Concomitant medications refer to all medications that started at any time and were taken at any time after the start of treatment until the end of the entire treatment period including those continued from pre-treatment.
- 3) Medications missing both start and stop dates, or having a start date prior to the last dose of study drug and missing the stop date, or having a stop date after the start of

study drug and missing the start date, will be counted as concomitant. When partial dates are present in the data, both a partial start date and/or a partial stop date will be evaluated to determine whether it can be conclusively established that the medication either ended prior to the start of study drug or started after the end of study drug. If the above cannot be conclusively established based on the partial and/or present dates, then the medication will be counted as concomitant.

# **6.2.3** Safety

1266

1267

1268

1269 1270

1271

1272

1273

12741275

1276

1277

- 1) If multiple results (e.g., lab test results) are reported at a study visit, then the last available result reported for that visit will be used in that visit summary.
- 2) Adverse events will be coded and classified using MedDRA. The specific dictionary version will be provided in the actual tables/listings.
- 3) Counting rules for AEs: AEs with missing start dates, but with stop dates either overlapping into the treatment period or missing, will be counted as treatment-emergent, taking the worst-case approach. Special care will be taken regarding partial dates with similar logic to that of the prior/concomitant medications applied.
- 4) For purposes of flagging individual subject data, laboratory test result abnormalities are defined as values above or below the normal range.
- 5) Conversion factor for temperature:
- Temperature (in  $^{\circ}$ C) = 5/9 (Temperature [in  $^{\circ}$ F]-32).
- 1279 Conversion factors for ECG QT to QTcF if any subjects do not have reported QTcF values but have reported QT and RR values:
- 1281 Fridericia formula:  $QTcF = QT / (RR^{1/3})$

#### 1282 **6.2.4** SAS® Procedures

- This section provides sample SAS<sup>®</sup> code to illustrate statistical tests specified in the statistical methods section. All computer output from SAS<sup>®</sup> statistical procedures serving as a basis for extracted results (e.g., MIXED, FREQ/CMH) will be retained for quality control procedures and will be included in CSR appendices.
  - 1) The percentage change from baseline is calculated as the post-baseline score minus the baseline score, and the difference divided by the baseline score, expressed in units of percent. The mean percentage change is derived as the least squares mean for treatment/visit interaction from the mixed model shown in 4) below.
  - 2) M-N Method:

The M-N method will be used for the primary efficacy analysis, which provides point estimates for the difference between treatments, and their corresponding

CONFIDENTIAL 50

12931294

1287

1288

1289

1290

1291

1292



























PASI is evaluated within each of the four body regions: a) head, b) upper limbs, c) trunk, and d) lower limbs;



1366

# APPENDIX 2 DLQI SCORING

The Dermatology Life Quality Index (DLQI) questionnaire is an assessment of treatment response on the subject's quality of life to measure how much the scalp psoriasis has affected the subject's life during the previous week.







